CLINICAL TRIAL: NCT04262518
Title: Feasibility of Integrating the Outcomes4Me Smartphone Navigation Application Into the Care Management of Breast Cancer Patients
Acronym: FIONA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Outcomes4Me (Industry)
Collaborators: Massachusetts General Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: O4M-B001
Record Dates: First submitted 2020-01-30; First posted 2020-02-10 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Breast Cancer; Invasive Breast Cancer; Metastatic Breast Cancer; Breast Carcinoma; Metastatic Breast Carcinoma
Keywords: Invasive Breast Cancer; Metastatic Breast Cancer; NCCN Guidelines; Patient Navigation; Treatment Options; Clinical Trial Options; Symptom Management
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Outcomes4Me App Users (Other): This cohort will download and use the Outcomes4Me mobile app for breast cancer.
  Interventions: Device: Outcomes4Me Mobile App

INTERVENTIONS:
Device: Outcomes4Me Mobile App — A mobile app that provides patient navigation and treatment and clinical trial options to people with breast cancer

SUMMARY:
This study aims to investigate the role of a mobile health app, Outcomes4Me, in the navigation of care for people with breast cancer.

DETAILED DESCRIPTION:
This protocol is a single arm pilot study of a novel breast cancer navigation app that is intended to assist patients with breast cancer understand their diagnosis and treatment options (both as part of standard of care practice and clinical trials) and manage their care, through treatment and symptom tracking. Patients will also be able to share information and get news via the app relevant to their cancer subtype. Results from this intervention will inform future clinical integration efforts, improve patient-centeredness of such an app-based health content and data platform, and inform the design of a larger, randomized study to demonstrate an improvement in patients' outcomes as well as enhanced Real-World Evidence (RWE) data collection.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older, with histologically or cytologically confirmed invasive breast cancer stage I-IV
* Must be on, or planning to be on within 4 weeks of registration, active therapy, with the intent to receive some element of active therapy > 28 days after registration
* Must be able to understand, read, and write in English and be able to sign informed consent
* Must have an Apple or Android smart phone that they are able to use and download the Outcomes4Me app on
* Must have the ability to access the internet at least once per week via their smart phone (having a computer is not required)

Exclusion Criteria:

* Participations seen for consultation opinion only and are not planning to receive some element of active treatment from an MGH medical or radiation oncology provider at MGH (Boston or Waltham sites) during the 12-week study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2020-08 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
Measure # of times a patient logs into the Outcomes4Me app over a 12 week period | 12 Weeks
  We will track engagement with the app by tracking the number of times a user logs in to the Outcomes4Me app over a 12 week period. The app will be considered feasible if at least 40% of enrolled patients engage with the Outcomes4Me app at least 3 times during the 12-week study period.

SECONDARY OUTCOMES:
Measure System-Usability Score (SUS) of app usage | 12 weeks
  Usability will be assessed using the System Usability Scale (SUS). We wil collect the input of breast cancer patients to the SUS questions, using in-app surveys and will calculate the SUS score. We will assess overall satisfaction with the app by asking users to provide an answer to the question "How likely are you to recommend this product to a friend" on a scale of 0-10.
Measure Net-Promoter Score (NPS) of app usage | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Maya Said, Sci.D, Study Chair — Outcomes4Me
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Isakoff SJ, Said MR, Kwak AH, Glieberman E, O'Rourke EA, Stroiney A, Spring LM, Moy B, Bardia A, Horick N, Peppercorn JM. Feasibility of introducing a smartphone navigation application into the care of breast cancer patients (The FIONA Study). Breast Cancer Res Treat. 2023 Jun;199(3):501-509. doi: 10.1007/s10549-023-06918-y. Epub 2023 Apr 27. PMID 37103597